CLINICAL TRIAL: NCT00492830
Title: A Phase 1, Open-label, Dose Escalation Study of the Humanized Monoclonal Antibody, TRC093, in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase 1, Open-label, Dose Escalation Study of TRC093, in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Bryan Leigh, MD, Medical Monitor, TRACON Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 093ST101
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Cancer; Neoplasm Metastasis
Keywords: Phase 1; TRC093; denatured collagen; solid tumor; antibody; TRACON; Locally advanced solid tumors; Metastatic solid tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TRC093 recombinant humanized IgG1k monoclonal antibody — TRC093 is a humanized monoclonal antibody to cleaved collagen administered i.v. on days 1 and 15 of each 28 day cycle until pregression or unacceptable toxicity develops.

SUMMARY:
This study is being performed to evaluate the safety and tolerability of the TRC093 antibody.

DETAILED DESCRIPTION:
In addition to safety, this study will also evaluate pharmacokinetics, tumor response, and anti-TRC093 antibody formation.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for study participation only if all of the following criteria apply:

1. The patient has given informed consent.
2. The patient is willing and able to abide by the protocol.
3. The patient is at least 18 years old.
4. The patient has advanced cancer and is not eligible for treatment or no effective treatment exists.
5. Significant toxicities resulting from prior therapy must have recovered.
6. If the patient is a female of childbearing potential, she is using an acceptable/effective method of contraception.
7. If the patient is a female, she has had a negative serum pregnancy test within the past 30 days.
8. The patient has adequate ability to perform activities of daily living.
9. The patient has adequate organ function as assessed by laboratory tests

Exclusion Criteria:

A patient will not be eligible for study participation if any of the following criteria apply:

1. The patient weighs more than 264 lbs.
2. The patient has had a major surgical procedure, or significant injury within the past 28 days or there is an anticipation of the need for major surgery during the course of the study.
3. The patient has received treatment for their cancer, including radiation (minimal amount of localized radiation may be allowed), within the past 28 days.
4. The patient has known brain tumors.
5. The patient experienced blood clots within six months prior to study start.
6. The patient has a non-healing wound, ulcer or bone fracture.
7. The patient received recent thrombolytic or anticoagulant therapy.
8. The patient has an unstable medical condition or significant comorbid pathophysiology (e.g. active infection, poorly controlled diabetes, unstable angina, severe heart failure) that would interfere with his/her participation in the study.
9. The patient enrolled, or plans to enroll, in a concurrent treatment protocol with another investigational product.
10. The patient is receiving, or plans to receive, an anti-cancer therapy during the study with the exception of patients receiving chronic luteinizing hormone-releasing hormone (LHRH) agonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated | Through last patient last visit
Dose Limiting Toxicities | 28 day evaluation period

SECONDARY OUTCOMES:
Pharmacokinetics of TRC093 monoclonal antibody | Through last patient last visit
Number of responses by tumor type | Through last patient last visit

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Santa Monica, California